CLINICAL TRIAL: NCT05814614
Title: Lower Urinary Tract Symptoms in Parkinson's Disease Effectiveness of Pelvic Floor Muscle Exercises and Electrical Stimulation, a Randomized Control Trial
Brief Title: Bladder Complaints in Parkinson's Disease Effectiveness of Pelvic Floor Muscle Exercises and Electrical Stimulation
Acronym: LIPPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Royal Dutch Society for Physical Therapy (Unknown); The Dutch Brain Foundation (Other)
Responsible Party: Principal Investigator, Dorien Bennink, Principal Investigator, clinical epidemiologist MSc, of the department of urology,, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL8301905822
Record Dates: First submitted 2022-12-14; First posted 2023-04-18 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Lower Urinary Tract Symptoms; Parkinson Disease
Keywords: Parkinson disease; Lower urinary tract symptoms; Electrical simulation; Pelvic floor muscle exercises; Bladder training; Biofeedback
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are assigned to three parallel arms for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electrical stimulation small phase duration (Active Comparator): phase duration 200 microseconds, frequency 20 Hertz, 20 minutes
  Interventions: Other: pelvic physical therapy
- electrical stimulation broad pulse duration (Active Comparator): phase duration 1000 microseconds, frequency 8 Hertz, 20 minutes
  Interventions: Other: pelvic physical therapy
- electrical stimulation inactive 100Hz (Sham Comparator): phase duration 200 microseconds, frequency 100 Hertz, 2 seconds active 20 seconds no output, 20 minutes
  Interventions: Other: pelvic physical therapy

INTERVENTIONS:
Other: pelvic physical therapy — Pelvic floor muscle exercises, biofeedback, bladder training

SUMMARY:
The goal of this clinical trial is to compare the effect of pelvic physical therapy with different types of electrical stimulation(ES) for bladder complaints in people with Parkinson's disease.

The main question it aims to answer is:

What is the effect of pelvic physical therapy with ES for bladder complaints in people with Parkinson's disease.

Secondary question:

What is the most effective type of ES on bladder complaints in people with Parkinson's disease.

Participants will be randomized into three groups. Two different kinds of ES and a sham group. Participants will receive eight session of pelvic physical therapy. Pelvic physical therapy consists of e.g. bladder training, pelvic floor muscle exercises and biofeedback.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common degenerative neurological disease in the elderly. PD is predominantly a movement disorder. In addition, PD is associated with non-motor and autonomic symptoms. Over 75% of PD patients, experience lower urinary tract symptoms (LUTS), one of the most common autonomic symptoms. LUTS consists of urgency, frequency and nocturia with or without urinary incontinence (UI). More than 60% of PD patients experience nocturia. LUTS have a negative impact on Quality of Life(QoL), increases the risk of falls are a barrier to exercise and may lead to early admission into care. Therefore, this potentially increases healthcare related costs. First treatment options for LUTS in the general population are conservative therapy and medication. Conservative therapy consists of e.g., behavioral advice, bladder training, pelvic floor muscle exercises provided by a pelvic physical therapist(PPT) and, electrical stimulation(ES). Knowledge of the effectiveness of conservative treatment options for LUTS in PD is limited. Although ES is used effectively in patients with LUTS, it has not yet been studied in PD patients. ES has hardly any side effects, but there is uncertainty about optimal ES parameters.

Objective: to study the effectiveness of pelvic physical therapy and ES in patients with PD suffering from LUTS.

Study design: Randomized Controlled Trial (RCT).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Questionnaires are online, allowing participants to complete the questionnaires at home at a convenient time.

Participants may have direct benefits of participating in this study. Participants included in the study will have two additional visits to a research PPT that will last one hour each, at baseline and after treatment. During this visit, a digital pelvic floor muscle (PFM) assessment and an EMG measurement of the PFM will be performed. EMG measurement will be done with a small anal- or vaginal probe. No risks are associated with the use of this probe.

Participants will be referred to local PPT's close to the subjects home address for the treatment sessions.

Intervention: eight treatment sessions of 30 minutes pelvic physical therapy over a 10-week period. The intervention consists of bladder- and behavioral advice, pelvic floor muscle exercises (PFME), urge suppression techniques, biofeedback and ES with an intra anal or intra vaginal probe. The group is divided into three groups. Group 1: ES with small pulse duration, group 2: ES with broad pulse duration, group 3: (control group) receiving sham ES.

No adverse events are expected since pelvic physical therapy and ES in LUTS is usual care in the general population in the Netherlands. Expected burden for the participants is very low.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease
* ≥ 18 years of age
* Self-reported LUTS
* Stable Parkinson's medication for at least three months
* Able and willing to independently read and fill in questionnaires in the Dutch language, sufficient understanding of Dutch language
* Able to independently visit a pelvic physical therapy practice

Exclusion Criteria:

* Patients with other neurological diseases
* Surgery in the pelvic region in the last year
* Cancer or cancer treatment in the pelvic region
* Pregnancy
* Current urinary tract infection
* Pure stress urinary incontinence without urgency, frequency, nocturia
* Botox, PTNS or pelvic physical therapy in the last year
* Sacral neuromodulator
* Pacemaker and Implantable cardioverter defibrillator (ICD)
* Deep Brain stimulation (DBS)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Change from baseline at 12 weeks
  Questionnaire of bladder function and urination, of last month, validated for men and
  women, 6-point-scale; contains 8 items, 3 about storage of urine, 4 about urination and 1 of quality of life.
  Total score of 0-35, with a minimal important difference(MID) of 3, validated in the Netherlands (MID 5.2) A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
  The IPSS is the most prevalent patient-administered questionnaire used in urology.

SECONDARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire-Urinary Incontinence Short form (ICIQ-UI SF) | Change from baseline at 12 weeks; at 24 weeks; at one year
  The validated ICIQ-UI SF measures frequency, severity and, impact on QoL in men and women. The ICIQ-UI SF consists of 4 questions on: frequency or urinary incontinence, amount of leakage, overall impact of urinary incontinence, self-diagnostic item. The score ranges between 0-21. A higher score represents worse QoL.
Change International Consultation on Incontinence Questionnaire-Lower Urinary Tract quality of life (ICIQ-LUTSqol) | Change from baseline at 12 weeks; at 24 weeks; at one year
  The validated ICIQ-LUTSqol measures QoL with particular reference to social effects.The ICIQ-LUTSqol consists of 20 questions. Total score ranges between 19-76 with greater values indicating increased impact on QoL. Bother scales are not incorporated in the overall score but indicate impact of individual symptoms for the patient.
Change in 24 hour bladder diary, bladder volume | Change from baseline at 12 weeks
  24 hour bladder diary: change in mean of bladder volume. Normal bladder volume ranges between: 250-500ml.
Change in 24 hour bladder diary, frequency of micturition | Change from baseline at 12 weeks
  24 hour bladder diary, change in frequency of micturition. Number of micturition's in 24 hours. Normal frequency with fluid intake of 1.5-2 liters is 6-8 times in 24 hour.
Change in 24 hour bladder diary, urgency | Change from baseline at 12 weeks
  24 hour bladder diary change in urgency scale: patient perception of intensity of urgency
  scale(PPIUS). 0 No urgency I felt no need to empty my bladder, but did so for other reasons.
  1. Mild urgency I could postpone voiding as long as necessary, without fear of wetting myself.
  2. Moderate urgency I could postpone voiding for a short while, without fear of wetting myself.
  3. Severe urgency I could not postpone voiding, but had to rush to the toilet in order not to wet myself.
  4. Urge incontinence I leaked before arriving to the toilet.
  A higher score on the PPIUS implicates more severe urgency complaints.
Change in 24 hour bladder diary, urinary incontinence | Change from baseline at 12 weeks
  24 hour bladder diary change in urinary incontinence episodes. Number of urinary incontinence episodes in 24 hours.
Change in International Prostate Symptom Score (IPSS) | Change from baseline at 24 weeks and at one year.
  Questionnaire of bladder function and urination, of last month, validated for men and women, 6-point-scale; contains 8 items, 3 about storage of urine, 4 about urination and 1 of quality of life.
  Total score of 0-35, with a minimal important difference(MID) of 3, validated in the Netherlands (MID 5.2).
  A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
  The IPSS is the most prevalent patient-administered questionnaire used in urology.
Change in International Consultation on Incontinence Questionnaire-Overactive Bladder Short form (ICIQ-OAB) | Change from baseline at 12 weeks; at 24 weeks; at one year
  The validated ICIQ-OAB evaluating overactive bladder and related impact on quality of life (QoL) and outcome of treatment in men and women, measure the impact of urinary frequency, urgency, urge incontinence and nocturia symptoms. It consist of 6 questions. The scores range from 0-16, overall score with greater values indicating increased symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Pelger, Prof., Study Chair — Head department urology Leiden University Medical Center
Locations (1):
- Leiden Univesity Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication. Data will be made (publicly) accessible following funder's guidelines, LUMC data management guidelines and following policies for availability of data, material and methods from publishers when submitting our manuscripts.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after publication of the results.
Access Criteria: Data can only be used for scientific research, not for educational purposes. Request will be reviewed by the research team.

REFERENCES:
- [Background] McDonald C, Rees J, Winge K, Newton JL, Burn DJ. Bladder training for urinary tract symptoms in Parkinson disease: A randomized controlled trial. Neurology. 2020 Mar 31;94(13):e1427-e1433. doi: 10.1212/WNL.0000000000008931. Epub 2020 Feb 13. PMID 32054791
- [Background] Sakakibara R, Panicker J, Finazzi-Agro E, Iacovelli V, Bruschini H; Parkinson's Disease Subcomittee, The Neurourology Promotion Committee in The International Continence Society. A guideline for the management of bladder dysfunction in Parkinson's disease and other gait disorders. Neurourol Urodyn. 2016 Jun;35(5):551-63. doi: 10.1002/nau.22764. Epub 2015 Mar 25. PMID 25810035
- [Background] Balash Y, Peretz C, Leibovich G, Herman T, Hausdorff JM, Giladi N. Falls in outpatients with Parkinson's disease: frequency, impact and identifying factors. J Neurol. 2005 Nov;252(11):1310-5. doi: 10.1007/s00415-005-0855-3. Epub 2005 May 18. PMID 15895303